CLINICAL TRIAL: NCT07231042
Title: Evaluation of Accuracy of Patient Specific Plate for Reduction and Fixation of Mandibular Angle Fracture
Brief Title: Evaluation of Accuracy of Patient-Specific Plate for Reduction and Fixation of Mandibular Angle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdulaziz Mohsen A Alanazi, Principal Investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TANTAOMFS-MAF-160
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mandibular Angle Fracture
Keywords: CAD/CAM; Patient-Specific Plate; Mandibular Fracture; Angle Fracture; Titanium Plate; Virtual Surgical Planning; Maxillofacial Trauma
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: A single-arm clinical study evaluating the accuracy, stability, and clinical outcomes of patient-specific titanium plates fabricated using CAD/CAM technology for fixation of mandibular angle fractures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient-Specific Titanium Plate Fixation (Experimental): All participants will undergo open reduction and internal fixation of displaced mandibular angle fractures using a patient-specific titanium plate fabricated by CAD/CAM technology. The customized plate provides accurate anatomical adaptation, enhanced stability, and reduced operative time.
  Interventions: Device: Patient-Specific Titanium Plate

INTERVENTIONS:
Device: Patient-Specific Titanium Plate — A customized titanium fixation plate designed using computer-aided design and manufacturing (CAD/CAM) technology based on preoperative CT data. The plate is fabricated to precisely match the patient's mandibular anatomy and used for open reduction and internal fixation of mandibular angle fractures.

SUMMARY:
This study evaluates the accuracy and clinical effectiveness of patient-specific titanium plates designed using CAD/CAM technology for the reduction and fixation of mandibular angle fractures. The customized plates are manufactured to match each patient's anatomical morphology, aiming to improve surgical precision, minimize operative time, and enhance postoperative stability. The study assesses clinical outcomes including pain, edema, occlusion, sensory recovery, maximal mouth opening, and radiographic bone healing across multiple follow-up periods. The goal is to determine whether patient-specific plates offer superior clinical and radiographic results compared with conventional fixation methods.

DETAILED DESCRIPTION:
This clinical study investigates the use of computer-aided design and computer-aided manufacturing (CAD/CAM) technology to fabricate patient-specific titanium plates for the reduction and fixation of mandibular angle fractures. The customized plates are created based on each patient's CT-derived anatomical morphology, allowing the surgical team to perform virtual planning, simulate fracture reduction, and generate an accurately fitted plate prior to surgery.

The primary objective of the study is to assess the accuracy of anatomical reduction achieved using patient-specific plates and to evaluate short- and medium-term clinical outcomes. All patients are treated using an intraoral surgical approach, with fracture reduction performed according to the preoperative virtual plan. The patient-specific titanium plate is then positioned and fixed without the need for intraoperative plate bending.

Clinical outcomes evaluated in this study include postoperative pain, facial edema, maximal mouth opening, sensory recovery of the inferior alveolar nerve, dental occlusion, and wound healing. Radiographic assessment evaluates bone healing, alignment, intergonial distance, and the accuracy of fracture reduction across multiple follow-up intervals. These evaluations aim to determine the stability and precision of the patient-specific fixation method.

The study follows patients through standardized follow-up periods, including immediate postoperative assessment, 1-week, 1-month, 3-month, and 6-month evaluations. Data are collected prospectively using unified clinical forms and radiological imaging protocols. All procedures adhere to ethical guidelines, and informed consent is obtained from all participants prior to enrollment.

The rationale behind using patient-specific plates is the potential to improve biomechanical stability, reduce operative time, eliminate intraoperative plate bending, and achieve more predictable postoperative outcomes. This study aims to provide evidence on whether CAD/CAM-based customized plates offer measurable advantages over conventional fixation systems in the treatment of mandibular angle fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with displaced mandibular angle fracture indicated for open reducation and internal fixation.
2. Age of patient > 18 years old .

Exclusion Criteria:

1- Medically compromised patients with impaired healing ability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Accuracy of Fracture Reduction | Immediately and 1 week postoperatively
  Accuracy of anatomical reduction will be evaluated by comparing postoperative CBCT scans with preoperative virtual surgical plans using superimposition analysis to measure the deviation between planned and achieved fragment positions.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | 1 day, 1 week, and 1 month postoperatively
  Pain intensity will be recorded using a Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst pain).
Postoperative Facial Edema | 1 week and 2 weeks postoperatively
  Facial swelling will be measured using the Souza JA facial edema scale based on standardized anthropometric landmarks.
Occlusal Relationship and Stability | 1 week, 1 month, and 3 months postoperatively
  Occlusal stability will be evaluated clinically using the Uglešić occlusion score to assess the degree of alignment and functional contact between opposing teeth
Recovery of Inferior Alveolar Nerve Function | 1 week, 1 month, and 3 months postoperatively
  Sensory recovery of the lower lip and chin will be assessed using light touch and two-point discrimination tests
Radiographic Bone Healing | 3 and 6 months postoperatively
  Bone union and callus formation will be assessed radiographically on CBCT images to confirm complete healing and stability at the fracture site.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulaziz M Alanazi, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Ibrahim M Nowair, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mona S sheta, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No